CLINICAL TRIAL: NCT07329855
Title: Analysis of Opioid Consumption After Thoracotomy and Factors Affecting Postoperative Acute Pain
Brief Title: Opioid Consumption After Thoracotomy and Factors Affecting Postoperative Acute Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Baldemir, Clinic Associate Professor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2024-KAEK-24/23
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Anesthesia; Thoracotomy; Opioid; Postoperative Pain Management; Length of Hospital Stay
Keywords: Thoracotomy; opioid consumption; postoperative acute pain; postoperative complications; length of hospital stay
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Analgesics, Opioid; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged over 18 years old scheduled for thoracotomy: The total intraoperative and postoperative opioid consumption will be determined. The effect of perioperative opioid use on postoperative acute pain, postoperative complications, and length of hospital stay will be investigated.
  Interventions: Other: Opioid Analgesic; Other: Pain Medicine

INTERVENTIONS:
Other: Opioid Analgesic — The total intraoperative and postoperative opioid consumption will be determined. The effect of perioperative opioid use on postoperative acute pain, postoperative complications, and length of hospital stay will be investigated.
Other: Pain Medicine — Pain levels of patients at 1, 2, 4, 8, 16, 24, and 48 hours after thoracotomy will be evaluated using the Visual Analog Scale (VAS).

SUMMARY:
Thoracic surgery operations constitute a significant portion of surgical procedures performed in hospitals. In the United States, more than 50,000 thoracic surgical procedures are performed annually, and more than 80% of these patients experience moderate to severe postoperative pain requiring opioid administration, which increases the risk of complications . It has also been reported that chronic pain develops in approximately 50% of patients after thoracic surgery .

Thoracic surgery is commonly associated with severe, multifactorial pain during the postoperative period and is among the surgical branches with a high risk of developing chronic pain Despite advances in understanding postoperative pain mechanisms and improvements in pain management, inadequate postoperative pain control remains an unresolved healthcare problem. Higher acute pain scores are associated with less effective ventilation and coughing, increased incidence of lower respiratory tract infections, and prolonged ICU and hospital stays .

In the management of acute postoperative pain after thoracic surgery, clinicians have sought alternatives to thoracic epidural analgesia to avoid its potential adverse effects. Truncal blocks such as thoracic paravertebral block, erector spinae plane block, and serratus anterior block have been used to reduce postoperative pain . Additionally, various other analgesic techniques such as patient-controlled analgesia (PCA) and multimodal analgesia have been employed. Historically, the cornerstone of acute postoperative pain control has been systemic opioids administered via oral, intravenous, or thoracic epidural routes . Although opioids provide excellent pain relief, they are associated with significant side effects that can adversely affect recovery .

With the increasing use of ultrasonography (USG), truncal blocks have become more widespread. Alongside the development of Enhanced Recovery After Thoracic Surgery (ERATS) protocols, efforts have been made to reduce opioid use, leading to differing opinions regarding the management of acute pain after thoracic surgery. To prevent opioid use disorder and potential side effects, opioid-free or opioid-sparing approaches are now being encouraged in perioperative pain management . Conversely, some studies suggest that intraoperative opioid administration may have favorable effects on postoperative acute and chronic pain. Previous research has reported that the average daily opioid consumption after thoracic surgery is approximately 30 morphine milligram equivalents (MME) .

Although video-assisted thoracoscopic surgery (VATS) has become more common, thoracotomy cases still constitute a large proportion of thoracic surgery procedures. Moreover, severe postoperative pain after thoracic surgery is most commonly associated with the thoracotomy incision itself. While some studies have suggested that new truncal block techniques may provide effective analgesia and reduce opioid consumption after thoracotomy, further studies are needed to determine which blocks are most commonly preferred and how opioid consumption patterns have changed with the adoption of these newer regional techniques.

A review of the current literature reveals that the factors influencing acute pain after thoracotomy have not been sufficiently evaluated. Therefore, a re-evaluation of the factors affecting acute pain following thoracotomy, considering recent developments in pain management, is necessary. Furthermore, examining the relationship between perioperative opioid consumption, postoperative complications, and hospital length of stay in this patient population will provide valuable contributions to the literature.

The aim of this study is to evaluate the amount of opioid consumption following thoracotomy and to investigate whether perioperative opioid use affects acute pain, postoperative complications, and the length of hospital stay.

DETAILED DESCRIPTION:
H₀ (Null Hypothesis):

Opioid consumption in patients after thoracotomy is not high (≤30 morphine milligram equivalents [MME]/day).

H₁ (Alternative Hypothesis):

Opioid consumption in patients after thoracotomy is high (>30 morphine milligram equivalents [MME]/day).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Patients scheduled for thoracotomy
* Patients with an American Society of Anesthesiologists (ASA) physical status classification of I-III
* Patients who have provided informed consent
* Patients with a body mass index (BMI) between 18-40 kg/m²

Exclusion Criteria:

* Patients with ASA class IV or higher
* Patients younger than 18 years old
* Patients with systemic inflammatory disease
* Patients receiving continuous anti-inflammatory and/or analgesic medication
* Patients with chronic preoperative pain
* Pregnant patients
* Outpatients who received anesthesia outside the operating room
* Emergency cases
* Patients who underwent VATS, sternotomy, mediastinoscopy, or tracheal resection
* Patients with a history of previous thoracic surgery
* Patients who had a thoracic epidural catheter inserted for postoperative pain management
* Patients with a BMI <18 or >40 kg/m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will begin prospectively and will be completed once the targeted number of patients has been reached. The study population will consist of patients over 18 years of age who are scheduled to undergo thoracotomy under general anesthesia at the operating rooms of the Department of Anesthesiology and Reanimation, University of Health Sciences, Ankara Atatürk Sanatorium Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | intraoperatively and for 24 hours postoperatively
Determination of the amount of opioid consumption after thoracotomy | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: ZİYA CAN KUŞ, Principal Investigator — ANKARA ATATURK SANATORİUM TRAİNİNG AND RESEARCH HOSPITAL
Locations (1):
- Ankara Ataturk Sanatorium Training and Research Hospital, Ankara, 06280, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No